CLINICAL TRIAL: NCT02584283
Title: A Multicenter Randomized Controlled Trial to Compare the Efficacy of End-ischemic Dual Hypothermic Oxygenated Perfusion With Standard Static Cold Storage of Liver Grafts Donated After Circulatory Death in Preventing Biliary Complications
Brief Title: Dual Hypothermic Oxygenated Perfusion of DCD Liver Grafts in Preventing Biliary Complications After Transplantation
Acronym: DHOPE-DCD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Robert J. Porte (Other)
Collaborators: Erasmus Medical Center (Other); Leiden University Medical Center (Other); Universitaire Ziekenhuizen KU Leuven (Other); University Hospital, Ghent (Other); King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor-Investigator, Robert J. Porte, Prof. dr., University Medical Center Groningen
Organization: University Medical Center Groningen (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DHOPE-DCD Trial
Record Dates: First submitted 2015-09-25; First posted 2015-10-22 (Estimated); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Liver Failure; End Stage Liver Disease; Biliary Tract Diseases
Keywords: Liver Transplantation; Donation after Circulatory Death; Machine Perfusion
MeSH Terms: conditions — Liver Failure; End Stage Liver Disease; Biliary Tract Diseases | interventions — newcastle organ perfusion fluid; Glutathione

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dual hypothermic oxygenated perfusion (Experimental): The liver is procured with a segment of supratruncal aorta. The intervention is restricted to the liver graft after arrival in the transplant center and before implantation. The donor liver is subjected to 2 hours of hypothermic oxygenated perfusion via the portal vein and the supratruncal aorta applied by the Liver Assist®. Before perfusion, the liver is flushed via the portal vein with 1 L Belzer machine perfusion solution. The perfusion is pressure controlled and set to a mean of 25 mmHg (arterial) and 5 mm Hg (portal). The perfusion fluid is 4 L Belzer machine perfusion solution with additional 3 mmol/L glutathione. The perfusion fluid is 12°C, when the temperature is set at 10°C. The oxygen flow is set at 0.5 mL/min of 100% oxygen on each of the two membrane oxygenators.
  Interventions: Procedure: Dual hypothermic oxygenated perfusion; Device: Liver Assist®; Procedure: Perfusion fluid; Drug: Glutathione
- Care as usual (No Intervention): The donor liver is procured with a segment of 5 cm circular supratruncal aorta left attached to the coeliac trunc. The patients randomized to the control group will receive a liver graft preserved by conventional SCS without any further intervention.

INTERVENTIONS:
Procedure: Dual hypothermic oxygenated perfusion — Dual hypothermic oxygenated perfusion using the Liver Assist
  Arms: Dual hypothermic oxygenated perfusion
Device: Liver Assist® — The Liver Assist® is the device used to give the intervention dual hypothermic perfusion.
  Arms: Dual hypothermic oxygenated perfusion
Procedure: Perfusion fluid — The perfusion fluid is Belzer machine perfusion solution University of Wisconsin (Bridge-to-Life, Ltd., Northbrook, IL).
  Arms: Dual hypothermic oxygenated perfusion
Drug: Glutathione — Glutathione in a dosage of 3 mmol/ is added to the perfusion fluid according to the intention of use of the perfusion fluid.
  Arms: Dual hypothermic oxygenated perfusion

SUMMARY:
Rationale: Recent publications report good results of controlled donation after circulatory death (DCD) Maastricht category III liver transplantation when strict donor-recipient matching is applied and ischemia times are kept to a minimum. However a major concern remains the high rate of biliary complications after transplantation of DCD livers. Non-anastomotic biliary strictures (NAS) occur in 29% of patients receiving a DCD graft whereas the incidence of NAS in recipients of donation after brain death (DBD) liver grafts is 11%. NAS are associated with higher morbidity and increased cost of liver transplantation. Injury to the biliary epithelium and the peribiliary vascular plexus occurring during donor warm ischemia and static cold storage (SCS) has been identified as a major risk factor for development of NAS. Machine perfusion has been proposed as an alternative strategy for organ preservation, offering the opportunity to improve the quality of the organ by providing oxygen to the graft. Experimental studies have shown that end-ischemic dual hypothermic oxygenated machine perfusion (DHOPE) helps liver grafts to recover from ischemia by restoring mitochondrial function. Moreover, DHOPE has been shown to provide better preservation of peribiliary vascular plexus of the bile ducts, which could be an important step forward in reducing the incidence of NAS after transplantation.

Objective: To study the efficacy of end-ischemic DHOPE in reducing the incidence of NAS within six months after controlled DCD (Maastricht category III) liver transplantation.

Study design: An international, multicenter, prospective, randomized, controlled, interventional, clinical trial with a two parallel arm approach (treatment/control).

Study population: Adult patients (≥18 yrs old) undergoing a liver transplantation with a liver graft procured from a controlled DCD donor (Maastricht category III) with a body weight ≥40 kg.

Intervention: In the intervention group liver grafts will be subjected to two hours of hypothermic, oxygenated perfusion at the end of SCS and before implantation. In the control group donor liver grafts will be preserved in accordance to standard practice by SCS only.

Main study parameters/endpoints: The incidence and severity of symptomatic NAS as diagnosed by an Adjudication committee (who are blinded for the group assignment) by means of magnetic resonance cholangiopancreatography (MRCP).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old)
* Signed informed consent
* Willing and able to attend follow-up examinations
* Donor liver graft from a controlled donation after circulatory death (Maastricht category III)
* Donors with a body weight ≥40 kg

Exclusion Criteria:

* Simultaneous participation in another clinical trial that might possibly influence this trial
* Mental conditions rendering the subject incapable to understand the nature, scope and consequences of the trial
* Listed for liver transplantation due to fulminant liver failure or retransplantation because of primary non-function
* Recipient positive test for HIV
* Donor positive for HIV antigen, hepatitis B core antibody, hepatitis B surface antigen, or hepatitis C antibody
* Simultaneous transplantation of another organ
* Patients with contra-indications for MRCP (i.e. pacemaker)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
The incidence of symptomatic non-anastomotic biliary strictures (NAS) | 6 months
  NAS is defined as all of the following criteria:
  * any irregularities or narrowing of the lumen of the intra- or extrahepatic donor bile ducts, but not at the anastomosis
  * which are diagnosed by cholangiogram (preferably by MRCP)
  * in the presence of a patent hepatic artery demonstrated by Doppler ultrasonography and if necessary, by computed tomography angiography
  * and as assessed by the Adjudication Committee
  * when imaging is indicated by clinical signs (i.e., jaundice, cholangitis) or elevation of cholestatic laboratory parameters in blood samples taken during follow-up

SECONDARY OUTCOMES:
Asymptomatic NAS | 6 months
  Asymptomatic NAS is defined as all of the following:
  * irregularities or narrowing of the lumen of the intra- or extrahepatic donor bile ducts, but not at the anastomosis
  * which are diagnosed by cholangiogram (preferably by MRCP)
  * in the presence of a patent hepatic artery demonstrated by Doppler ultrasonography and if necessary, by computed tomography angiography
  * in the absence of clinical signs (i.e., jaundice, cholangitis) or elevation of cholestatic laboratory parameters in blood samples taken during follow-up
The severity of NAS | 6 months
  Severity and location of NAS is based on assessment of the images of the MRCP obtained in all patients at six months after transplantation (time window of 15 days) which will be performed based on a scoring system described by Buis et. al. And required treatment for NAS (i.e. ursodeoxycholic acid, ERCP, retransplantation)
The location of NAS | 6 months
  Assessment of the images of the MRCP obtained in all patients at six months after transplantation (time window of 15 days) which will be performed based on a scoring system described by Buis et. al.
Graft (censored and uncensored for patient death) survival | 7 days, 1, 3 , 6, and 12 months after transplantation
Patient survival | 7 days, 1, 3 , 6, and 12 months after transplantation
Primary non-function | 7 days
  Defined as liver failure requiring retransplantation or leading to death within seven days after transplantation without any identifiable cause such as surgical problems, hepatic artery thrombosis, portal vein thrombosis and acute rejection
Initial poor function | 7 days
  Defined as a modification of the Olthoff criteria: Prothrombin time/ international normalized ratio (INR) >1.6 and or serum total bilirubin >10 mg/dL on postoperative day 7
Biochemical analysis of graft function and ischemia-reperfusion injury | Postoperative day 0 - 7 and 1, 3, 6 months
  serum levels of alanine aminotransferase (ALT), AST, alkaline phosphatase (AlkP), gamma-glutamyl transferase (γGT), and total bilirubin
Blood pressure | 5 min before reperfusion, at reperfusion and after 10 and 20 minutes of reperfusion
  mm Hg
Heart rate | 5 min before reperfusion, at reperfusion and after 10 and 20 minutes of reperfusion
  beats per minute
Vasopressor dosage | 5 min before reperfusion, at reperfusion and after 10 and 20 minutes of reperfusion
  microgram/kg/min
Length of stay | 6 months
  Length of initial ICU and initial hospital stay is determined in days of admission following liver transplantation. Duration of follow-up hospital stay is determined in days of hospital admission after discharge and up to six months after liver transplantation
Postoperative complications | 6 months
  According to the comprehensive complication index (CCI)
Renal function | day 7, and 1, 3, 6 months
  Estimated glomerular filtration rate (eGFR) according to the 4-variable Modification of Diet in Renal Disease (MDRD) equation
Flow | At 0, 15, 30, 45, 60, 75, 90, 105, 120 minutes after start of perfusion
  ml/min
Pressure | At 0, 15, 30, 45, 60, 75, 90, 105, 120 minutes after start of perfusion
  mm Hg
Resistance | At 0, 15, 30, 45, 60, 75, 90, 105, 120 minutes after start of perfusion
  ml/min/mm Hg
(In selected centers) value of perfusate's pH | At 5 minutes before and at 0.5 hour, 1 hour, 1.5 hours and 2 hours after start of perfusion
(In selected centers) value of perfusate's sodium | At 5 minutes before and at 0.5 hour, 1 hour, 1.5 hours and 2 hours after start of perfusion
  mmol/L
(In selected centers) value of perfusate's potassium | At 5 minutes before and at 0.5 hour, 1 hour, 1.5 hours and 2 hours after start of perfusion
  mmol/L
(In selected centers) value of perfusate's bicarbonate | At 5 minutes before and at 0.5 hour, 1 hour, 1.5 hours and 2 hours after start of perfusion
  mmol/l
(In selected centers) value of perfusate's lactate | At 5 minutes before and at 0.5 hour, 1 hour, 1.5 hours and 2 hours after start of perfusion
  mmol/l
(In selected centers) value of perfusate's alanine transaminase (ALT) | At 5 minutes before and at 0.5 hour, 1 hour, 1.5 hours and 2 hours after start of perfusion
  U/L
(In selected centers) value of perfusate's aspartate transaminase (AST) | At 5 minutes before and at 0.5 hour, 1 hour, 1.5 hours and 2 hours after start of perfusion
  U/L
(In selected centers) value of perfusate's alkaline phosphatase (AlkP) | At 5 minutes before and at 0.5 hour, 1 hour, 1.5 hours and 2 hours after start of perfusion
  U/L
(In selected centers) value of perfusate's gamma glutamyltransferase (γGT) | At 5 minutes before and at 0.5 hour, 1 hour, 1.5 hours and 2 hours after start of perfusion
  U/L
(In selected centers) value of perfusate's urea | At 5 minutes before and at 0.5 hour, 1 hour, 1.5 hours and 2 hours after start of perfusion
  mmol/L
(In selected centers) value of perfusate's total bilirubin | At 5 minutes before and at 0.5 hour, 1 hour, 1.5 hours and 2 hours after start of perfusion
  umol/l
(In selected centers) value of perfusate's thrombomodulin | At 5 minutes before and at 0.5 hour, 1 hour, 1.5 hours and 2 hours after start of perfusion
  pg/dl
(In selected centers) value of perfusate's high mobility group box-1 (HMBG) protein | At 5 minutes before and at 0.5 hour, 1 hour, 1.5 hours and 2 hours after start of perfusion
  μg/mL
(In selected centers) value of perfusate's cytochrome C | At 5 minutes before and at 0.5 hour, 1 hour, 1.5 hours and 2 hours after start of perfusion
(In selected centers) level of miRNA CDmiR-30e in perfusate | At 5 minutes before and at 0.5 hour, 1 hour, 1.5 hours and 2 hours after start of perfusion
  relative levels compared to perfusate
(In selected centers) level of miRNA CDmiR-222 in perfusate | At 5 minutes before and at 0.5 hour, 1 hour, 1.5 hours and 2 hours after start of perfusion
  relative levels compared to perfusate
(In selected centers) level of miRNA CDmiR-296 in perfusate | At 5 minutes before and at 0.5 hour, 1 hour, 1.5 hours and 2 hours after start of perfusion
  relative levels compared to perfusate
(In selected centers) level of miRNA HDmiR-122 in perfusate | At 5 minutes before and at 0.5 hour, 1 hour, 1.5 hours and 2 hours after start of perfusion
  relative levels compared to perfusate
(In selected centers) level of miRNA HDmiR-148a in perfusate | At 5 minutes before and at 0.5 hour, 1 hour, 1.5 hours and 2 hours after start of perfusion
  relative levels compared to perfusate
Histopathological status liver and bile ducts (in selected centers) | Within 0 to 30 minutes before perfusion, at 2 hours of perfusion, and at 1 hour after reperfusion
New onset diabetes after transplantation | 90 days
  * Symptoms of diabetes and random plasma glucose ≥11.1 mmol/L. Symptoms include polyuria, polydipsia, and unexplained weight loss. OR
  * Fasting plasma glucose ≥7.0 mmol/L. Fasting is defined as no caloric intake for at least eight hours. OR
  * Two-hour plasma glucose ≥11.1 mmol/L during an oral glucose tolerance test. The test should be performed as described by the WHO, using a glucose load containing the equivalent of 75 g anhydrous glucose dissolved in water.
Costs of treatment (in selected centers) | within 6 months after transplantation, including transplant operation
  according to the Cost and Outcome analysis of Liver Transplantation (COLT) study
Health related quality of life | within 6 months before transplantation and 6 months after transplantation
  EQ6D questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Porte, MD PhD Prof, Principal Investigator — University Medical Center Groningen
Locations (6):
- Belgium (2):
  - Ghent University Hospital, Ghent, De Pintelaan 185
  - University Hospitals Leuven, Leuven, Herestraat 49
- Netherlands (3):
  - Leiden Universtiy Medical Center, Leiden, South Holland
  - University Medical Center Groningen, Groningen
  - Erasmus Medical Center, Rotterdam
- King's College Hospital NHS Trust, London, United Kingdom

REFERENCES:
- [Derived] van Rijn R, Endo C, Kucukerbil EH, Blokzijl H, Blondeel J, Cortes Cerisuelo M, Coenraad MJ, Darwish Murad S, Doukas M, Eker H, de Haas RJ, Huurman VAL, de Meijer VE, Monbaliu D, Schurink IJ, Slangen JJG, Polak WG, de Jonge J, Porte RJ. Long-term Follow-up After Hypothermic Oxygenated Machine Perfusion in DCD Liver Transplantation: Results of a Randomized Controlled Multicenter Trial (DHOPE-DCD). Ann Surg. 2025 Nov 1;282(5):717-724. doi: 10.1097/SLA.0000000000006876. Epub 2025 Aug 5. PMID 41082480
- [Derived] Endo C, van Rijn R, Huurman V, Schurink I, van den Berg A, Murad SD, van Hoek B, de Meijer VE, de Jonge J, van der Hilst CS, Porte RJ. Cost-effectiveness of Dual Hypothermic Oxygenated Machine Perfusion Versus Static Cold Storage in DCD Liver Transplantation. Transplantation. 2025 Feb 1;109(2):e101-e108. doi: 10.1097/TP.0000000000005232. Epub 2024 Oct 8. PMID 39853733
- [Derived] van Rijn R, Schurink IJ, de Vries Y, van den Berg AP, Cortes Cerisuelo M, Darwish Murad S, Erdmann JI, Gilbo N, de Haas RJ, Heaton N, van Hoek B, Huurman VAL, Jochmans I, van Leeuwen OB, de Meijer VE, Monbaliu D, Polak WG, Slangen JJG, Troisi RI, Vanlander A, de Jonge J, Porte RJ; DHOPE-DCD Trial Investigators. Hypothermic Machine Perfusion in Liver Transplantation - A Randomized Trial. N Engl J Med. 2021 Apr 15;384(15):1391-1401. doi: 10.1056/NEJMoa2031532. Epub 2021 Feb 24. PMID 33626248
- [Derived] de Vries Y, Berendsen TA, Fujiyoshi M, van den Berg AP, Blokzijl H, de Boer MT, van der Heide F, de Kleine RHJ, van Leeuwen OB, Matton APM, Werner MJM, Lisman T, de Meijer VE, Porte R. Transplantation of high-risk donor livers after resuscitation and viability assessment using a combined protocol of oxygenated hypothermic, rewarming and normothermic machine perfusion: study protocol for a prospective, single-arm study (DHOPE-COR-NMP trial). BMJ Open. 2019 Aug 15;9(8):e028596. doi: 10.1136/bmjopen-2018-028596. PMID 31420387
- [Derived] van Rijn R, van den Berg AP, Erdmann JI, Heaton N, van Hoek B, de Jonge J, Leuvenink HGD, Mahesh SVK, Mertens S, Monbaliu D, Muiesan P, Perera MTPR, Polak WG, Rogiers X, Troisi RI, de Vries Y, Porte RJ. Study protocol for a multicenter randomized controlled trial to compare the efficacy of end-ischemic dual hypothermic oxygenated machine perfusion with static cold storage in preventing non-anastomotic biliary strictures after transplantation of liver grafts donated after circulatory death: DHOPE-DCD trial. BMC Gastroenterol. 2019 Mar 12;19(1):40. doi: 10.1186/s12876-019-0956-6. PMID 30866837